CLINICAL TRIAL: NCT05494905
Title: Effect of Virtual Reality and Functional Strength Training on Arm Function in Children With Cerebral Palsy_2021
Brief Title: Virtual Reality vs Functional Strength Training in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgia State University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Yuping Chen, Professor, Georgia State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: H21384
Record Dates: First submitted 2022-08-03; First posted 2022-08-10 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Virtual Reality; Functional Strength Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: For the first six weeks of intervention, children will be randomly assigned to receive either VR or FST. After being determined as a respondent or non-respondent by the end of the first 6 weeks of the intervention, non-respondent children will be re-randomized to either receive the combination of FST and VR or switch to the other intervention (i.e., children who receive VR in the first 6 weeks will switch to FST; and verse versa).
Who Masked: Outcomes Assessor
Masking Description: The therapist who conducts the assessments will be blinded with the intervention these children receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) (Experimental)
  Interventions: Other: VR
- Functional Strength Training (FST) (Active Comparator)
  Interventions: Other: FST

INTERVENTIONS:
Other: VR — In this project, the investigators focus on using our developed VR gaming platform called Super Pop VR, a VR system that can be individualized to the movement capabilities of the child. It consists of the Microsoft Kinect camera, a laptop, software, and TV screen. The research team will loan the system to the family. While engaged with the game, the child is immersed in a virtual world where virtual objects appear on the screen surrounding the child. Children are asked to move their arms to 'pop' as many virtual objects as possible in a certain amount of time. Playstation 2 EyeToy and EyeToy 2 games will also be used to increase children's motivation by playing a variety of different VR games.
  Arms: Virtual Reality (VR)
Other: FST — FST involves repetitive progressive resistance exercise during goal-directed functional activity with the children focus on the activity being performed. Children will be offered a pamphlet containing suggested functional arm exercises and these exercises are designed to move the more affected arm in overhead, outward, and across midline directions. Each exercise will be embedded in a game-like activity. Children will start with no resistance and gradually add on resistance using elastic bands or weight cuffs.
  Arms: Functional Strength Training (FST)

SUMMARY:
Virtual reality (VR) has shown to be effective to improve arm function in children with cerebral palsy (CP). Recently, functional strength training (FST) starts to show to improve arm function in patients with stroke but has not been extensively explored in children with CP. This pilot study is to examine the effect of FST and VR on improving arm function in children with CP using a sequential multiple assignment randomized trial (SMART) to develop valid, high-quality adaptive intervention using VR and FST to improve arm function in children with CP. There is a growing interest and need for research on how to adapt and re-adapt intervention in children with CP in order to maximize clinical benefits. The treatment adapted here is by augmenting or switching to the other intervention.

Forty children with spastic type of CP will be recruited from the greater Atlanta area. Children will be randomly assigned to receive either VR or FST for 6 weeks (60 minutes per day, 3 days per week). After receiving 6 weeks of intervention, the children will be evaluated to determine whether they are responders or non-responders. For those who are responders, they will continue receiving the same dosage and type of intervention. That is, children who are assigned to VR will continue receiving VR for the next 6 weeks; children who are assigned to FST will continue receiving FST for the next 6 weeks. For those who are non-responders, children will be randomly assigned to augmenting the other intervention or switching to the other intervention. That is, for children who are assigned to augmenting the other intervention (i.e. the combination group), they will receive the combination of FST and VR for the next 6 weeks. For children who are assigned to switch to the other intervention, children who are assigned to VR in the first 6 weeks will receive FST for the next 6 weeks; whereas children who are assigned to FST in the first 6 weeks will receive VR for the next 6 weeks. Similar instruction, visit, and email reminder will be conducted as what they receive in the first 6 weeks. At the end of the study, children and primary caregivers will be interviewed to understand their perception about the intervention they have received.

The research team is expected children with CP will improve their arm function regardless which intervention they are assigned; however, children received VR will have a better improvement in arm function as compared with those who received FST at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* children are between ages 5-17 years
* diagnosed with CP;
* have a Manual ability classification system (MACs) level I-III;
* able to sit with trunk supported;
* are able to reach forward for more than half of their arm length;
* are able to comprehend a 3-step command;
* are able to see video screen (with or without corrected vision); and
* their primary caregiver is willing to follow the desired intervention 'dosing' and all evaluation measurements.

Exclusion Criteria:

* children have received surgery or botulinum toxin type A injection in the training arm within the preceding 4 months or are scheduled to receive it during the planned study period,
* if children have a severe attention deficit or uncontrolled epilepsy which may possibly be triggered by the light or sound of the video games.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reaching kinematics at the baseline | At baseline
  Reaching kinematics will be assessed while the child is interacting with Super Pop VRTM, wherein virtual bubbles are projected onto the TV in randomly dispersed locations, using the Kinect system. Three testing bubbles will be tested in the location where children need to reach about arm length overhead at 180, 135, and 90 degrees of shoulder abduction, with instructions for children to reach in two conditions: 1) as fast as possible, and 2) as accurate as possible. Position data from the Kinect will be converted into 3-dimensional coordinate data and kinematic variables (movement time, trajectory straightness, speed, smoothness) will be computed.
Reaching kinematics at the end of the 6th week | The end of the 6th week
  Reaching kinematics will be assessed while the child is interacting with Super Pop VRTM, wherein virtual bubbles are projected onto the TV in randomly dispersed locations, using the Kinect system. Three testing bubbles will be tested in the location where children need to reach about arm length overhead at 180, 135, and 90 degrees of shoulder abduction, with instructions for children to reach in two conditions: 1) as fast as possible, and 2) as accurate as possible. Position data from the Kinect will be converted into 3-dimensional coordinate data and kinematic variables (movement time, trajectory straightness, speed, smoothness) will be computed.
Reaching kinematics at the end of the 12th week | The end of the 12th week
  Reaching kinematics will be assessed while the child is interacting with Super Pop VRTM, wherein virtual bubbles are projected onto the TV in randomly dispersed locations, using the Kinect system. Three testing bubbles will be tested in the location where children need to reach about arm length overhead at 180, 135, and 90 degrees of shoulder abduction, with instructions for children to reach in two conditions: 1) as fast as possible, and 2) as accurate as possible. Position data from the Kinect will be converted into 3-dimensional coordinate data and kinematic variables (movement time, trajectory straightness, speed, smoothness) will be computed.
Fine motor domain of Peabody Developmental Motor Scales-2nd edition at baseline | At baseline
Fine motor domain of Peabody Developmental Motor Scales-2nd edition at the end of the 6th week | The end of the 6th week
Fine motor domain of Peabody Developmental Motor Scales-2nd edition at the end of the 12th week | The end of the 12th week
Daily use of affected hand at baseline | At baseline
  Daily use of affected hand will be evaluated using Revised Pediatric Motor Activity Log (R-PMAL), which is filled by primary caregivers about how often and how well their children use the affected arm in daily activities.
Daily use of affected hand at the end of the 6th week | The end of the 6th week
  Daily use of affected hand will be evaluated using Revised Pediatric Motor Activity Log (R-PMAL), which is filled by primary caregivers about how often and how well their children use the affected arm in daily activities.
Daily use of affected hand at the end of the 12th week | The end of the 12th week
  Daily use of affected hand will be evaluated using Revised Pediatric Motor Activity Log (R-PMAL), which is filled by primary caregivers about how often and how well their children use the affected arm in daily activities.

SECONDARY OUTCOMES:
Muscle strength at baseline | At baseline
  Muscle strength of shoulder flexion, extension, abductor, adduction, external rotation, and international rotation, elbow flexion and extension, and wrist flexion and extension will be measured using hand-held dynamometer prior and after intervention.
Muscle strength at the end of the 6th week | The end of the 6th week
  Muscle strength of shoulder flexion, extension, abductor, adduction, external rotation, and international rotation, elbow flexion and extension, and wrist flexion and extension will be measured using hand-held dynamometer prior and after intervention.
Muscle strength at the end of the 12th week | The end of the 12th week
  Muscle strength of shoulder flexion, extension, abductor, adduction, external rotation, and international rotation, elbow flexion and extension, and wrist flexion and extension will be measured using hand-held dynamometer prior and after intervention.
Children's motivation and compliance | During the 12 weeks of intervention
  Children's motivation and compliance to the intervention will also be evaluated using the daily activity training log. The primary caregiver will be asked to keep an activity training log to record their child's training activity, including the daily training and the total time when the child takes part in the training. The total duration of performing the VR or conventional program will be calculated as the measure of compliance. The investigators will ask caregivers to record the reasons for not completing the daily training.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Chen, ScD, PT, Principal Investigator — Department of Physical Therapy, Georgia State University
Locations (1):
- Department of Physical Therapy, Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No